CLINICAL TRIAL: NCT02996344
Title: Suicide Prevention Training for Primary Care Providers-in-training
Brief Title: Suicide Prevention Training for PC Providers-in-training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Wendi Cross, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00061161
Record Dates: First submitted 2016-10-24; First posted 2016-12-19 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Didactic training (Active Comparator): Behavioral; participants will view the approximately one hour Commitment to Living: Primary Care (CTL:PC) didactic training videos.
  Interventions: Other: Didactic training
- Didactics and standardized patients (Experimental): Behavioral; participants will view the approximately one hour Commitment to Living: Primary Care (CTL:PC) didactic training videos plus two practice standardized patient interactions.
  Interventions: Other: Didactic training; Other: Standardized patient interaction

INTERVENTIONS:
Other: Didactic training — Six online training modules pertaining to suicide prevention in primary care.
Other: Standardized patient interaction — Two standardized patient practice interactions - 1 face-to-face, 1 remote/telehealth.
  Arms: Didactics and standardized patients

SUMMARY:
This randomized control study responds to the need for effective suicide prevention education/training that is grounded in adult learning theory and advances in education, in the context of a changing health care landscape where primary care providers are likely to encounter suicidal individuals. The study will test the effectiveness of suicide prevention education for providers-in-training by comparing two conditions: 1) A Control learning group: includes suicide prevention didactics (Commitment to Living: Primary Care) delivered online via brief videos, and 2) An Experimental learning group: includes didactics plus two standardized patient (SP) interactions. One Experimental learning group SP interaction will be in person and the other will be conducted remotely using a secure webcam service (OoVoo). All SP interactions will be recorded. Both groups will be compared in terms of their suicide prevention skills using an SP 'test case' at 6-month follow up. The primary research question is to learn about the impact of practice (though SP simulation) over and above didactics alone.

DETAILED DESCRIPTION:
Suicide is a national public health crisis and a critical patient safety issue. Suicide is the 10th leading cause of death overall and, shockingly, the 2nd leading cause of death in adolescents and young adults (15-34 years old). 1 A recent U.S. study of suicide reported that 45% of individuals who died by suicide had contact with primary care services within one month before their death. 2 Another study found that 80% of youth who died by suicide saw their primary care provider within the year of their death. 3 Patient safety is compromised when primary care providers lack the knowledge and skills to assess and respond to patients at risk for suicide.

This randomized control study responds to the need for effective suicide prevention education/training that is grounded in adult learning theory and advances in education, in the context of a changing health care landscape where primary care providers are likely to encounter suicidal individuals. 4 We will test the effectiveness of suicide prevention education for providers-in-training by comparing two conditions: 1) A Control learning group: includes suicide prevention didactics (Commitment to Living: Primary Care) delivered online via brief videos, and 2) An Experimental learning group: includes didactics plus two standardized patient (SP) interactions. One Experimental learning group SP interaction will be in person and the other will be conducted remotely using a secure webcam service (OoVoo). All SP interactions will be recorded. Both groups will be compared in terms of their suicide prevention skills using an SP 'test case' at 6-month follow up. The primary research question is to learn about the impact of practice (though SP simulation) over and above didactics alone. The hypotheses are as follows:

H1: All subjects will demonstrate improved suicide prevention knowledge from pre to post didactics and maintain improvement 6 months after didactics.

H2: Subjects in the experimental learning group will report greater satisfaction with the training, greater self-efficacy in identifying and responding to patients at risk for suicide, greater intention to use, as well as use of suicide prevention skills.

H3: Subjects in the experimental learning group will also be more skillful in responding to patients at risk for suicide (in an SP interview, measured by objective observed ratings) compared to the control learning group 6 months after didactics.

Exploratory Aims: We will examine moderators of outcomes, differences among SP simulations (i.e., face-to-face vs. telehealth modalities), and if there is growth in improved skills observed over multiple SP experiences in the experimental learning group.

ELIGIBILITY:
Inclusion Criteria:

* trainee in family medicine residency, pediatrics residency, or nurse practitioner program at URMC.
* speaks/writes English.

Exclusion Criteria:

* on academic probation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Mean score using the Commitment to Living: Primary Care Observational Rating form | through study completion, an average of 6 months
  Each participant will be evaluated via standardized patient interactions which are video taped and reliably coded using the Commitment to Living: Primary Care Observational Rating form. Score will range from 0 - 32.

SECONDARY OUTCOMES:
Changes in suicide prevention knowledge | 1 day following enrollment and 15 days from enrollment
  Participants will complete a 17-item knowledge questionnaire prior to and following the online didactic training. Number of correct responses will be compared.
Changes in suicide prevention self-efficacy | 1 day following enrollment and 15 days from enrollment
  Participants will complete a 20-item 5-point likert scale self-efficacy questionnaire prior to and following the online didactic training. Average responses will be compared.
Changes in suicide prevention knowledge | 15 days from enrollment and through study completion, an average of 6 months
  Participants will complete a 17-item knowledge questionnaire following the online didactic training and end of study. Number of correct responses will be compared.
Number of participants intending to transfer training to practice | 15 days from enrollment and through study completion, an average of 6 months
  Participants will complete a 8-item intentions to use training in practice on a 5-item likert scale questionnaire following the online didactic training and end of study. Number of participants who report positive intentions to use the training in practice will be compared.
Changes in suicide prevention self-efficacy | 15 days from enrollment and through study completion, an average of 6 months
  Participants will complete a 20-item 5-point likert scale self-efficacy questionnaire following the online didactic training and end of study. Average responses will be compared.
Use of suicide prevention skills | through study completion, an average of 6 months
  Participants will self-report whether they used suicide prevention skills in practice on 0-4 point likert scale, with 0 defined as no use and 4 as frequently used.
Feedback on training | through study completion, an average of 6 months
  Participants will provide feedback on their experience with suicide prevention training on 15 items using a 5-point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Wendi F Cross, PhD, Principal Investigator — Associate Professor of Psychiatry (Psychology) and Pediatrics
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmedani BK, Simon GE, Stewart C, Beck A, Waitzfelder BE, Rossom R, Lynch F, Owen-Smith A, Hunkeler EM, Whiteside U, Operskalski BH, Coffey MJ, Solberg LI. Health care contacts in the year before suicide death. J Gen Intern Med. 2014 Jun;29(6):870-7. doi: 10.1007/s11606-014-2767-3. Epub 2014 Feb 25. PMID 24567199
- [Background] Bridge JA, Horowitz LM, Fontanella CA, Grupp-Phelan J, Campo JV. Prioritizing research to reduce youth suicide and suicidal behavior. Am J Prev Med. 2014 Sep;47(3 Suppl 2):S229-34. doi: 10.1016/j.amepre.2014.06.001. PMID 25145744
- [Background] Wyzga RE. The effect of air pollution upon mortality: a consideration of distributed lag models. J Am Stat Assoc. 1978;73(363):463-72. doi: 10.1080/01621459.1978.10480035. No abstract available. PMID 12262745
- [Background] Pisani AR, Cross WF, Watts A, Conner K. Evaluation of the Commitment to Living (CTL) curriculum: a 3-hour training for mental health professionals to address suicide risk. Crisis. 2012 Jan 1;33(1):30-8. doi: 10.1027/0227-5910/a000099. PMID 21940243
- [Background] Aiken LS, West SG. Multiple regression: Testing and interpreting interactions. Newbury Park, CA: Sage; 1991.
- [Derived] Cross WF, West JC, Pisani AR, Crean HF, Nielsen JL, Kay AH, Caine ED. A randomized controlled trial of suicide prevention training for primary care providers: a study protocol. BMC Med Educ. 2019 Feb 14;19(1):58. doi: 10.1186/s12909-019-1482-5. PMID 30764814